CLINICAL TRIAL: NCT06939569
Title: A Bidirectional, Multicenter Cohort Study of Inflammatory Bowel Disease (IBD) Patients With Nonalcoholic Fatty Liver Disease (NAFLD)
Brief Title: An Observational Study of Inflammatory Bowel Disease (IBD) Patients With Non-alcoholic Fatty Liver Disease (NAFLD)
Status: Recruiting | Type: Observational
Sponsor: Shanghai East Hospital (Other)
Collaborators: Shanghai Pudong New Area Health Commission (Unknown); Dongfang Hospital Affiliated to Tongji University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-PWDL-01
Record Dates: First submitted 2025-04-20; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Inflammatory Bowel Disease (IBD); Metabolic Dysfunction Associated Fatty Liver Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IBD with MASLD

SUMMARY:
Inflammatory bowel diseases (IBD), including ulcerative colitis and Crohn's disease, are currently of unknown etiology and incurable. In recent years, the incidence of IBD has increased dramatically in China, and it will become a common disease of digestive system in China. Mesenteric adipose tissue hyperplasia indicates disease activity in IBD patients, and abnormal lipid metabolism plays an important role in the pathogenesis of IBD.

In addition to intestinal symptoms, nonalcoholic fatty liver disease (NAFLD), also known as metabolic dysfunction associated fatty liver disease (MASLD), has become the most common extraintinal manifestation in IBD patients. What are the similarities and differences between IBD patients with and without MASLD? Does the occurrence and severity of MASLD affect the clinical efficacy of IBD and increase the adverse outcome of IBD? There are no relevant studies to date. We have previously completed the construction of a cohort of 290 IBD patients using the IBD patient database and biobank of Dongfang Hospital, based on which we completed a cohort study on the effect of small intestinal bacterial overgrowth on IBD disease activity. Based on this cohort, multi-center cooperation was carried out to establish an IBD research cohort by collecting basic clinical information and biological samples such as peripheral blood and intestinal mucosa. The clinical characteristics of IBD patients with MASLD were analyzed. logistic regression, COX regression, Kaplan-Meier survival curve and other methods were used. To investigate the effect of MASLD on the clinical efficacy and prognosis of inflammatory bowel disease (IBD). This project will provide efficient, full and reliable research-grade data with Chinese characteristics for IBD clinical research, and improve the level of regional diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged over 18 years (including borderline values), of either sex.
2. Subjects consistented with the Chinese consensus on the diagnosis and treatment of IBD;
3. Subjects able to cooperate with follow-up, participate in this study and sign the informed consent.

Exclusion Criteria:

1. Subjects with incomplete clinical data;
2. Subjects can not to cooperate with follow-up, and refuse to sign the informed consent;
3. Subjects can not to cooperate with the completion of relevant examinations; 4 Pregnant women;

5.Subjects with severe heart, lung, kidney and other organ diseases or cancer, and expected survival time less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with IBD by imaging, histology and/or endoscopy in IBD Diagnosis and Treatment Center of East Hospital, Pudong New Area, Shanghai
Sampling Method: Non-Probability Sample
Enrollment: 337 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical remission or Endoscopic remission | Follow-up for 54 weeks
  Clinical remission (CDAI≤150 in CD patients, Mayo≤2 in UC patients); Endoscopic remission (SES-CD in CD patients and UCEIS in UC patients with > 50% improvement from baseline)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No